CLINICAL TRIAL: NCT00800917
Title: A Phase II Study of Temsirolimus and Bevacizumab in Recurrent Glioblastoma Multiforme
Brief Title: A Study of Temsirolimus and Bevacizumab in Recurrent Glioblastoma Multiforme
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: University of Copenhagen (Other); Wyeth is now a wholly owned subsidiary of Pfizer (Industry); Roche, Copenhagen (Unknown)
Responsible Party: Ulrik Lassen, MD, PH.D., Rigshospitalet
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BEV-CCI-779-GBM-02; Eudract no.: 2008-003679-40
Record Dates: First submitted 2008-12-01; First posted 2008-12-02 (Estimated); Last update posted 2010-06-02 (Estimated); Status verified 2010-04

CONDITIONS: Glioblastoma Multiforme
MeSH Terms: conditions — Glioblastoma | interventions — temsirolimus; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Temsirolimus — 25 mg weekly IV
Drug: Bevacizumab — 10 mg/kg every 2 weeks

SUMMARY:
This trial is an investigator initiated, open label phase II study, where patient with recurrent primary GBM will be considered for the study. Only patients with recurrence after Temozolomide and VEGF-directed therapy with Bevacizumab will be considered for the study. Patients will receive temsirolimus 25 mg IV over 30-60 minutes on days 1, 8, 15 and 22 and bevacizumab 10 mg/kg IV over 30-90 minutes on day 8 and 22. Treatment repeats every 28 days for a maximum of 12 courses in the absence of disease progression or unacceptable toxicity. A safety analysis will be performed when the first 10 patients have received minimum 4 cycles (8 weeks). The study will then be stopped:

If DLT is observed in > 2/10 patients, Occurrence of any serious adverse events not described in the SPC of each agents, If partial remission is not observed in at least 1/10 patients

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Histological verification of primary GBM and failure after radiotherapy and temozolomide (TMZ)
* Previously treated with VEGF-directed therapy with bevacizumab
* Previously received radiotherapy and temozolomide
* More than 4 weeks since any of the following prior treatments: chemotherapy (6 weeks for nitrosoureas or mitomycin C)
* Radiotherapy to nontarget lesions or lesions that are not to be biopsied VEGF-directed therapy (including bevacizumab)
* Investigational agents
* More than 6 months since prior major surgery or open biopsy and recovered (only 6 weeks required if operation is for recurrent GBM)
* No concurrent medications or substances known to affect or with the potential to affect the activity or pharmacokinetics of the following:

  * Temsirolimus
  * Bevacizumab
  * CYP450 isoenzymes
  * ECOG performance status 0-1
  * WBC ≥ 3,000 mm³
  * Absolute neutrophil count ≥ 1,500/mm³
  * Platelet count ≥ 100,000/mm³
  * Bilirubin and phosphate normal
  * AST and ALT ≤ 2.5 times upper limit of normal
  * Creatinine normal OR creatinine clearance ≥ 60 mL/min
  * Urine protein: creatinine ratio < 1.0 OR 24-hour urine protein < 1,000 mg
  * Fasting cholesterol < 350 mg/dL (cholesterol medications are allowed)
  * Fasting triglycerides < 400 mg/dL
  * PT INR ≤ 1.5
  * Hematocrit < 41% (for males) or < 38% (for females)
  * Fertile females must use an approved contraceptive (p-pills, IUD, depot injection of gestagen, subdermal implantation, hormonal vaginal ring or transdermal depot plaster), throughout the study and 3 months after discontinuation of study drugs. Fertile men must use dobbelt barrier method (preservative with sperm inhibiting creme) or female partner uses the above mentioned contraceptive.
* Fertile males must use preservatives.

Exclusion Criteria:

* Clinically significant cardiovascular disease, including the following:
* Cerebrovascular accident within the past 6 months
* Transient ischemic attack within the past 6 months
* Myocardial ischemia within the past 6 months
* Myocardial infarction within the past 6 months
* Other thromboembolic event within the past 6 months
* Unstable angina within the past 6 months
* Uncontrolled hypertension (i.e., hypertension despite maximal therapy)
* New York Heart Association class II-IV heart disease
* Congestive heart failure
* Serious cardiac arrhythmia requiring medication
* Clinically significant peripheral vascular disease
* Uncontrolled intercurrent illness
* Ongoing or active infection
* One of the following within the past 6 months
* Abdominal fistula
* Gastrointestinal perforation
* Intra-abdominal abscess
* Serious or nonhealing wound, ulcer, or bone fracture
* Psychiatric illness or social situations that would preclude study compliance
* Uncontrolled diabetes
* Hemoglobin A1c > 7%
* Concurrent non-study related surgical procedures
* Concurrent treatment with CYP3A4 inducers or inhibitors
* Other concurrent anticancer agents or therapies
* Significant traumatic injury within the past 28 days
* History of allergic reactions to compounds of similar chemical or biological composition to temsirolimus or bevacizumab
* Hypersensitivity to Chinese hamster ovary cell products or other recombinant human antibodies (e.g., infliximab)
* Pregnancy or nursing
* Patients previously intolerant to bevacizumab
* Anticoagulant therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2008-11; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Progression-free survival in months | From start of treatment to death or progression

SECONDARY OUTCOMES:
Adverse events | every 2 weeks
Objective tumor response rate | every 8 weeks
Pre- vs post-treatment measurements of biomarkers and vascular system/immune system parameters | weekly for the first 4 weeks, then every 8 weeks
Correlation with biomarkers | at the end of the study

CONTACTS AND LOCATIONS:
Locations (1):
- Rigshospitalet, Copenhagen, Denmark